CLINICAL TRIAL: NCT02080546
Title: Vaginal Cuff Dehiscence and Thermal Injury at the Time of Total Laparoscopic Hysterectomy: A Review of the Duke Experience and Randomized Controlled Trial
Brief Title: Vaginal Cuff Dehiscence and Thermal Injury During TLH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00019452
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-01

CONDITIONS: Vaginal Cuff Dehiscence; Thermal Injury
Keywords: Vaginal cuff dehiscence; Thermal Injury; Total laparoscopic hysterectomy

ARMS (2):
- Cut/Coag (Active Comparator)
  Interventions: Procedure: Cut-Coag; Device: Valleylab G3000 Electrosurgical Device
- V-mode (Experimental)
  Interventions: Procedure: V-mode; Device: Valleylab G3000 Electrosurgical Device

INTERVENTIONS:
Procedure: Cut-Coag — Incision using electrothermal cautery, with an attempt made to use the "cut" (continuous low-voltage, high-current) for colpotomy incision following the initial scoring of the cervico-vaginal tissue on the "coag" (pulsed high-voltage, low-current) mode.
  Other Names: Valleylab G3000 Electrosurgical Device
  Arms: Cut/Coag
Procedure: V-mode — Incision using electrothermal cautery in the "V mode". The V mode combines real-time tissue sensing technology with the cut and coag waveforms to reduce the amount of thermal spread to the tissue without sacrificing hemostasis during monopolar electrothermal procedures.
  Other Names: Valleylab G3000 Electrosurgical Device
  Arms: V-mode
Device: Valleylab G3000 Electrosurgical Device — Use of surgical device Valleylab G3000 Electrosurgical Device

SUMMARY:
Purpose of this randomized control study is to determine if the mode of electrothermal colpotomy incision affects (1) the degree of thermal injury at the time of laparoscopic hysterectomy or (2) the incidence of clinical surrogates of compromised vaginal cuff healing. Women already scheduled for TLH will be randomized to colpotomy incision with the V mode or standard cut/coag form of electrothermal energy.

Prevalence of vaginal cuff injury will be calculated, and cross tabulation tables will be used to examine the association fo dehiscence with proposed risk factors in the retrospective part of the study. In the randomized controlled trial, depth of thermal injury will be compared between the two groups, and a chi-square test will be used to test for a difference in clinical outcomes between the two groups. There is little risk associated with this study above the normal surgical risks; however, the V mode has not been previously been studied for its use in making a colpotomy incision. Loss of confidentiality is a risk of the study, but all samples will be de-identified and given a unique study number, and only individuals directly involved in the study will be given access to the study information.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patient scheduled for total laparoscopic hysterectomy (TLH)
3. Signed informed consent

Exclusion Criteria:

1. Known pelvic infection within 30 days prior to hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-12; Primary Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula S Lee, MD, Principal Investigator — Duke University

REFERENCES:
- [Derived] Teoh D, Lowery WJ, Jiang X, Ehrisman J, Halvorson P, Broadwater G, Bentley R, Secord AA, Sobolewski C, Berchuck A, Havrilesky LJ, Valea FA, Lee PS. Vaginal cuff thermal injury by mode of colpotomy at total laparoscopic hysterectomy: a randomized clinical trial. J Minim Invasive Gynecol. 2015 Feb;22(2):227-33. doi: 10.1016/j.jmig.2014.10.002. Epub 2014 Oct 8. PMID 25305572

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 subjects either withdrew or were excluded from the study. Thermal injury could not be assessed in 18 specimens because of sampling error.
Period: Overall Study
Arm/Group | Cut/Coag | V-mode
Started | 57 | 63
Completed | 49 | 52
Not Completed | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cut/Coag | V-mode | Total
Number analyzed (Participants) | 49 | 52 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 43 | 79
  >=65 years | 13 | 9 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12.5) | 54 (11.9) | 56.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 52 | 101
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 48 | 51 | 99
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 14 | 23
  White | 39 | 36 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 52 | 101
Body Mass Index [Median (Full Range); unit: kg/m^2] | 33 [20 to 54] | 32 [20 to 50] | 32.5 [20 to 54]

OUTCOME MEASURES:

1. Primary Outcome: Degree of Thermal Injury at the Time of Laparoscopic Hysterectomy
Description: distance in millimeters over which thermal tissue injury extends (henceforth referred to as "injury").
Time Frame: up to 36 months
Population: 49 participants were included in the cut/coag arm and 52 participants in the V mode arm. Thermal injury was assessed at the anterior margin in 91 specimens and at the posterior margin in 93 specimens.
Measure: Mean (Full Range); unit: mm
Units Other Than Participants: Vaginal Cuff Specimens
Arm/Group | Cut/Coag | V-mode
Number analyzed (Participants) | 44 | 49
Number analyzed (Vaginal Cuff Specimens) | 87 | 97
mm
  Anterior Depth of thermal injury (mm) | 0.68 [0.18 to 1.43] | 0.63 [0.3 to 1.4]
  Posterior Depth of thermal injury (mm) | 0.66 [0.15 to 1.55] | 0.70 [0.2 to 1.63]

2. Secondary Outcome: Incidence of Clinical Surrogates of Compromised Vaginal Cuff Healing
Description: a difference between arms in the proportion of patients who have at least one of the following post-operatively: vaginal vault granulation tissue, vaginal cuff separation/dehiscence, or vaginal apex infection
Time Frame: 4 weeks, 3 months, and 6 months after hysterectomy for a post-operative check and pelvic examination
Population: This secondary objective was not evaluated
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Cut/Coag | V-mode
Number analyzed (Participants) | 49 | 52
participants
  Granulation Tissue 4 weeks post-op | 6 [1 to 11] | 8 [2 to 20]
  Granulation Tissue 3 months post-op | 18 [8 to 34] | 21 [9 to 36]
  Granulation Tissue 6 months post-op | 10 [2 to 27] | 11 [2 to 28]
  Vaginal cuff induration 4 weeks post-op | 2 [0 to 11] | 4 [0 to 14]
  Vaginal cuff induration 3 months post-op | 0 [0 to 0] | 5 [1 to 17]
  Vaginal cuff induration 6 months post-op | 0 [0 to 0] | 0 [0 to 0]
  Vaginal cuff infection 4 weeks post-op | 4 [0 to 14] | 0 [0 to 0]
  Vaginal cuff infection 3 months post-op | 0 [0 to 0] | 10 [3 to 24]
  Vaginal cuff infection 6 months post-op | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cut/Coag | V-mode
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/52
Other Adverse Events (participants affected / at risk) | 0/49 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes